CLINICAL TRIAL: NCT05617170
Title: The Role of Early Rehabilitation in Improving Stroke Systems of Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohmed Alaa Eldeine Ahmed, The Role of early rehabilitation in improving Stroke systems of Care, Assiut University
Other Study IDs: 123456789
Record Dates: First submitted 2022-10-16; First posted 2022-11-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-12

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group 1 experimental group will subject to implanted rehabilitation programme: 50 case of acute cerebrovascular stroke patients will subject to implanted rehabilitation programme based on telemedicine if avilable .
  Interventions: Other: Rehabilitation
- Group 2 control group will subject to ordinary rehabilitation techniques: 50 control patients of acute cerebrovascular stroke patients will subject to ordinary rehabilitation techniques .
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — 50 case of acute cerebrovascular stroke patients will subject to implanted early rehabilitation programme based on telemedicine if avilable .
  50 control patients of acute cerebrovascular stroke patients will subject to ordinary rehabilitation techniques .

SUMMARY:
1. To assess the effect of implementing stroke early rehabilitation using telemedicine if avialable in the stroke unit of the Neurology Department , Assuit university hospitalis , Egypt.
2. Importance and impact of this programme on function and quality of life after stroke

DETAILED DESCRIPTION:
In this case control study,we will analyzed Patients admitted to Neurology Depatment in assuit university hospitals from 1/2023 until 1/2024 and divide them in two groups , Group receive early rehabilitation services with the personnel get tele-rehab training and the other group get training with the usual pathway in the hospital by other personnel, and we could follow up the two groups for 3 months and comparing both groups .

ELIGIBILITY:
Inclusion Criteria:

1. Mild to Moderate stroke Patients (ischemic or hemorrhagic) admitted to AUH within 24 hour after admission.
2. ALL age Groups .
3. Both Sex.
4. Group receive rehab services with the personnel get tele-rehab training and the other group get training with the usual pathway in the hospital by other personnel, and we could follow up the two groups for 3 months and comparing both groups .

Exclusion Criteria:

Severe Stroke.

* Stroke Mimmics .
* Pregnancy.
* Stroke with severe hepatic ,renal and Pulmonary diseases limiting or affecting early rehabilitation .

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * 50 case of acute cerebrovascular stroke patients will subject to implanted programme of early rehabilitation based on Telemedicine .
  * 50 control Patient of acute cerebrovascular stroke will subject to ordinary rehabilitaion techniques .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
• To assess the effect of implementing stroke early rehabilitation using telemedicine if avilable in the stroke unit of the Neurology Department , Assuit university hospitalis , Egypt. | 2 years
  In this case control study,we will analyzed Patients admitted to Neurology Depatment in assuit university hospitals from 1/2023 until 1/2024 and divide them in two groups , Group receive rehab services with the personnel get tele-rehab training and the other group get training with the usual pathway in the hospital by other personnel, and we could follow up the two groups for 3 months and comparing both groups .
  And we will analyize the effect of implanted programme on patients with cerebrovascular stroke .

CONTACTS AND LOCATIONS:
Overall Officials: Mohmed Ahmed, Proffessor, Principal Investigator — Faculty of Medicine , Assuit University , Egypt

IPD SHARING:
Plan to Share IPD: No